CLINICAL TRIAL: NCT02193659
Title: Changes Induced by Breakfast Cereals Enriched With Omega-3 in the Lipidic Profile: a Randomized Simple Controlled Trial
Brief Title: Changes Induced by Breakfast Cereals Enriched With Omega-3 in the Lipidic Profile
Acronym: cereals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Elena García García, PhD, PID, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Elena García-García 3; Enrique Roche Collado (Other Grant/Funding Number: Instituto de Salud Carlos III-FEDER PS09/01093)
Record Dates: First submitted 2014-02-23; First posted 2014-07-17 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Overweight
Keywords: breakfast cereal; omega-3; cholesterol; lipidic profile; consumption; acceptability
MeSH Terms: conditions — Overweight | interventions — Edible Grain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cereals (Experimental): For 30 days, participants in group 1 took cereals with omega-3 in the breakfast with diet, group 2 took cereals and diet, and group 3 only received the diet. The energy intake of the designed diet was similar into the three groups (ranging 1900-2000 Kcal per day).
  Interventions: Dietary Supplement: Cereals

INTERVENTIONS:
Dietary Supplement: Cereals — The participants were randomly single blind controlled trial distributed into three groups: (1, n =38), (2, n =38), (3, n =37). For 30 days, participants in group 1 took cereals with omega-3 in the breakfast with diet, group 2 took cereals and diet, and group 3 only received the diet.
  Other Names: Papilla multicereales con Omega-3 0628413; Papilla multicereales 0528413

SUMMARY:
The inclusion of breakfast cereals enriched with omega-3 for female users of a pharmacy who had some lipidic profiles to the limit is highly conditioned by their nutritional acceptance. The main objective is to assess the effect of breakfast cereals intake with omega-3 on women lipid profile values to the limit, users of a pharmacy in Elche and in this way reduce the small dyslipidemia.

DETAILED DESCRIPTION:
The investigators performed an intervention including 133 women (age 25-70 years). Participants were randomly and single-blind distributed into three groups: Group 1 (n=38) consumed cereal with omega-3 (Cw-3 + D), cereal (C) and diet (D), Group 2 (n=38). Volunteers consumed (C) + (D) and Group 3 (n=37) consumed only diet. All groups followed a limit levels-cholesterol diet. Circulating total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and glucose were determined at the beginning and end of a 30-day test.

Statistical analysis was carried out using STATGRAPHICS Centurion XV software (StatPoint Technologies, Inc. Warrington, VA, USA); likewise, significance was defined at p ≤ 0.05. Data are reported as mean ± standard error of the mean (sem). Intra-group statistical comparisons were performed using the following hypothesis tests, both parametric and non-parametric: t-test, sign test and signed rank test for paired samples. Inter-group statistical comparisons were performed using the one-way analysis of variance and the Kruskal-Wallis hypothesis tests. Also, Fisher's least significant difference (LSD) Multiple Range Test and Tukey's honestly significant difference (HSD) were used in order to determine which means were significantly different from the others. In addition, Generalized Multiple Regression was used to statistically analyze the relationships between the variations in the lipid profile and the different factors included in the study.

ELIGIBILITY:
Inclusion Criteria:

* voluntarily participation
* ages between 25-70 years
* undergoing dyslipidemia
* with no pharmacological treatment
* cholesterol (250-300 mg/dL)
* triglycerides (160-175 mg/dL)

Exclusion Criteria:

* subjects undergoing any pharmacological treatment that may influence lipid metabolism
* lipid levels outside the range of those specified in the inclusion criteria
* subjects that were deemed to be unlikely to complete the treatment or to cooperate fully at the investigator´s discretion.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Cholesterol Total characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  Circulating parameters of cholesterol total

SECONDARY OUTCOMES:
Weight (Kg) of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table the investigators present the weight of the three intervented groups
Cholesterol HDL characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  Circulating parameters of cholesterol HDL
Cholesterol LDL characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  Circulating parameters of cholesterol LDL
Triglycerides characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  Circulating parameters of triglycerides
Glucose characteristics of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  Circulating parameters of glucose
BMI (Kg/m2) of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table the investigators present the BMI of the three intervented groups
Hip/waist measure (cm) of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table the investigators present the hip / waist measure of the three intervented groups
Systolic pressure (mmHg) of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table the investigators present the systolic pressure of the three intervented groups
Diastolic pressure (mmHg) of volunteers at the beginning (day 1) and at the end of the study (day 30). Data are mean ± sem. | 30 days
  In this table the investigators present the diastolic pressure of the three intervented groups

CONTACTS AND LOCATIONS:
Overall Officials: Elena García-García, PDI, Principal Investigator — Universidad Miguel Hernandez de Elche
Locations (1):
- Pharmacy Iborra Campos, Elche, Alicante, Spain